CLINICAL TRIAL: NCT03299296
Title: Thromboprophylaxis in Patients Undergoing Orthopedic Surgeries; Focus on Cost-effective Analysis and Safety Comparison Between Rivaroxaban and Enoxaparin
Brief Title: Thromboprophylaxis in Patients Undergoing Orthopedic Surgeries; Comparison Between Rivaroxaban and Enoxaparin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ahmed AbdelMoneim Hassan Ali (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Sponsor-Investigator, Ahmed AbdelMoneim Hassan Ali, Assistant Lecturer of Clinical Pharmacy, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: FW A00015574
Record Dates: First submitted 2017-09-19; First posted 2017-10-03 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Thromboses, Deep Vein; Surgery--Complications
Keywords: Thromboprophylaxis; orthopedic; rivaroxaban; enoxaparin
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: single blind, sequentially simple randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban arm (Experimental): Rivaroxaban 10 Milligrams
  Interventions: Drug: Rivaroxaban 10 Milligrams
- Enoxaparin Arm (Active Comparator): 'Enoxaparin 40 Milligrams /0.4 Milliliters Prefilled Syringe
  Interventions: Drug: Enoxaparin 40 Milligrams/0.4 Milliliters Prefilled Syringe

INTERVENTIONS:
Drug: Rivaroxaban 10 Milligrams — The first group is to be on Rivaroxaban 10 mg with dosage according to the orthopedic approved regimen (10 mg once daily 6-10 hours after the surgery; recommended total duration of therapy: 12 to 14 days; The American College of Chest Physicians (ACCP) recommendation: Minimum of 10 to 14 days; extended duration of up to 35 days suggested.
  Arms: Rivaroxaban arm
Drug: Enoxaparin 40 Milligrams/0.4 Milliliters Prefilled Syringe — The other group will be administered the standard of care (SOC) enoxaparin as follows:
  Once-daily dosing: 40 mg once daily, with initial dose within 9 to 15 hours before surgery, and daily for at least 10 days (or up to 35 days postoperatively) or until risk of deep venous thrombosis (DVT) has diminished or the patient is adequately anticoagulated on warfarin. The American College of Chest Physicians recommends initiation ≥12 hours preoperatively or ≥12 hours postoperatively; extended duration of up to 35 days suggested.
  Arms: Enoxaparin Arm

SUMMARY:
The main objective is to reduce the incidence of venous thromboembolism (VTE) in orthopedic postoperative patients based on the potential benefit of using rivaroxaban as a monotherapy.

It is around efficacy and safety evaluation of using rivaroxaban as a monotherapy prophylactic agent in patients undergoing orthopedic surgeries taking into the account the reliable selection of patients most benefit.

Answering questions about additional cost benefit from the perceptive of the cost-effective analysis on extrapolating the results emerged to our university teaching hospital setting are going to be evaluating as well.

DETAILED DESCRIPTION:
There is a Today consensus that patients undergoing high-risk surgery should receive prophylaxis against postoperative venous thromboembolism (VTE). A good example of that could be orthopedic surgeries which place patients at unnecessary increased risk of fatal pulmonary embolism. For many years, pharmacotherapy options have been recommended by the American College of Chest Physicians (ACCP) for postoperative thromboprophylaxis were low-molecular-weight heparins (LMWHs), fondaparinux, and warfarin. However, their limitations have been repeatedly demonstrated in a huge number of randomized controlled trials (RCTs).

Since its introduction, low-molecular-weight heparins (LMWHs) are still common used in practice as thromboprophylactic agent. But, they require subcutaneous administration which making it challenging for use in settings other than the inpatient one. Despite the lower incidence of low-molecular-weight heparins (LMWHs) induced heparin-induced thrombocytopenia (HIT) compared with unfractionated heparins (UFH) in the postoperative setting, the risk of LMWH induced HIT in patients treated for VTE still concerns many clinicians. In addition to its subcutaneous administration, fondaparinux is contraindicated in severe renal impairment patients (with creatinine clearance (CrCl) <30 milliliter/minute) and those who have low body weight (<50 kg; venous thromboembolism prophylaxis only). While available orally, Vitamin K antagonists (VKAs) like Warfarin have unpredictable pharmacologic effects requiring a wakeful monitoring. Warfarin is also a remarkable source of food and drug interactions. As a result, it is mandatory to search for novel drugs or at least to search for new indications of really existing drugs.

In July 2011, the Food and Drug Administration (FDA) approved an orally administered selective factor Xa inhibitor called Rivaroxaban for the prevention of deep vein thrombosis (DVT) after total hip replacement (THR) or total knee replacement (TKR) surgeries. According to the Regulation of Coagulation in Orthopedic Surgery to Prevent Deep Vein Thrombosis and Pulmonary Embolism (RECORD) trials, rivaroxaban demonstrated superiority to enoxaparin in reducing venous thromboembolism without significant increase of bleeding risk. Rivaroxaban is recommended to be used at a fixed dose of 10 mg daily, with or without food, for 35 days following THR or 12 days following TKR.

Although the US Food and Drug Administration (FDA) advisory committee has recommended approval of rivaroxaban, many questions have been raised on the Regulation of Coagulation in Orthopedic Surgery to Prevent Deep Vein Thrombosis and Pulmonary Embolism (RECORD) trials of rivaroxaban. Some may argue that dosing was inconsistent with the recommendations. Others went far to say that the duration of treatment was inconsistent and did vary with enoxaparin. In other words, it was somewhat short.

Results from the ORTHO-TEP registry on joint replacement arthroplasty (hip and knee) from Dresden, Germany and Xarelto® in the Prophylaxis of Postsurgical Venous Thromboembolism after Elective Major Orthopaedic Surgery of the Hip or Knee (XAMOS) study are in accordance with the conclusion of Regulation of Coagulation in Major Orthopedic surgery reducing the Risk of DVT and PE (RECORD) trials. A subset of countries that participated in XAMOS also included patients undergoing fracture-related orthopedic surgery.

Moreover, very few randomized clinical trials (RCTs) are powered to study side effects when comparing substances, and even large RCTs may be too small to reveal rare side effects. It seems difficult to compare safety data from trial to trial because there is no standardized definition of bleeding. One prospective study collecting data from the electronic health record at two institutions concluded that using of enoxaparin for venous thromboembolism prophylaxis following total hip arthroplasty (THA) and total knee arthroplasty (TKA) was associated with a lower rate of the primary outcome (any postoperative bleeding) compared with the use of rivaroxaban in a similar cohort of patients. However, it was a retrospective investigation with many limitations can be argued with regard to selection and change in practice guideline during the study period.

Finally, there is lack of literature data that define rivaroxaban as orthopedic postoperative thromboprophylactic agent rather than well-known indications (hip and knee replacements). It also is not plausible to accurately compare safety data with other injectable anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

1. Undergo Orthopedic Surgery
2. Thromboprophylaxis Decision Taken
3. At least 18 years of age

Exclusion Criteria:

1. Planned intermittent pneumatic compression
2. A requirement for anticoagulant therapy that could not be stopped
3. Severe hypersensitivity reaction (eg, anaphylaxis) to rivaroxaban or enoxaparin.
4. Received another anticoagulant for more than 24 hours
5. Active bleeding or a high risk of bleeding
6. Thrombocytopenia associated with a positive test for antiplatelet antibody.
7. Warfarin associated international normalized ratio (INR) more than 1.5 on the day of the surgery
8. Conditions preventing bilateral venography
9. Intensive care unit (ICU) stay after surgery
10. Pregnant or breast-feeding
11. Creatinine clearance less than 30 ml per minute or acute renal failure before the surgery or at any point during the study period.
12. Moderate or Severe (Child Pugh B or C) hepatic Impairment or in patients with any hepatic disease associated with coagulopathy.
13. Concomitant use of drugs that are both P--glycoprotein inhibitors and moderate to strong cyp3a4 (ketoconazole, itraconazole, lopinavir/ritonavir, ritonavir, indinavir/ritonavir & conivaptan)
14. Creatinine clearance (CrCl) 15 to 80 mL/min and concurrent use of P-glycoprotein inhibitors or moderate CYP3A4 inhibitors (eg, abiraterone acetate, diltiazem, dronedarone, erythromycin, verapamil)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Any deep-vein thrombosis (DVT) | up to 35 days
  Validated clinical prediction rule like Wells Clinical Model is recommended to estimate pretest probability of deep venous thrombosis. Duplex ultrasonography is the preferred test to diagnose deep-vein thrombosis (DVT).
  Symptoms and signs of DVT may include unilateral leg swelling, pain in the affected leg, calf tenderness in affected leg, increased leg warmth, erythema of affected leg, or a "palpable cord" may be felt in the affected leg.
  DVT is going to be assessed using Clinical assessment, D-dimer test, Duplex ultrasonography and Venography according to Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines and based on availability and clinical circumstances.
Nonfatal pulmonary embolism (PE) | up to 35 days
  Regarding Pulmonary Embolism (PE), diagnosis is suspected in patients with dyspnea, tachypnea, pleuritic chest pain, cough, and/or fever. Diagnosis begins with initial risk stratification "Wells Clinical Model for Evaluating the Pretest Probability of pulmonary embolism (PE) " based on presence of shock or persistent hypotension to identify patients at high risk of early mortality.
  PE is going to be assessed using Clinical assessment, D-dimer test, Computerized tomography, Ventilation/perfusion (V/Q) scanning and Pulmonary angiography according to American College of Chest Physicians Evidence-Based Clinical Practice Guidelines and based on availability and clinical circumstances.
Death | up to 35 days
  Death from any cause including venous thromboembolism

OTHER OUTCOMES:
Major bleeding risk | After 4 hours of the first dose and up to 2 days after the last dose of the study drug.
  The incidence of major bleeding beginning after the first dose of the study drug and up to 2 days after the last dose of the study drug (on-treatment period). Major bleeding is defined as bleeding that is fatal, occurs in a critical organ (e.g., retroperitoneal, intracranial, intraocular, and intraspinal bleeding), or requires reoperation or extra surgical-site bleeding that was clinically overt and is associated with a fall in the hemoglobin level of at least 2 g per deciliter or that requires transfusion of 2 or more units of whole blood or packed cells.
Other on-treatment bleeding | After 4 hours of the first dose and up to 2 days after the last dose of the study drug.
  These include any on-treatment non major bleeding, hemorrhagic wound complications (a composite of excessive wound hematoma and reported surgical-site bleeding), and any bleeding that starts after the first oral dose of rivaroxaban and ended up to 2 days after the last dose is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AH Hassan Ali, master, Principal Investigator — School of Pharmacy Beni Suef University

IPD SHARING:
Plan to Share IPD: Yes
I'm going to share individual participant data with the ethical committee upon request for validation of research conduct at any time and after the finish of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within the study period and after finishing it.
Access Criteria: upon any request from Faculty of Medicine Beni Suef University Research Ethical Committee at any time of the study period, the hard cover of any documented will be delivered by hand to the Chairperson of the committee

REFERENCES:
- [Background] Beyer-Westendorf J, Lutzner J, Donath L, Tittl L, Knoth H, Radke OC, Kuhlisch E, Stange T, Hartmann A, Gunther KP, Weiss N, Werth S. Efficacy and safety of thromboprophylaxis with low-molecular-weight heparin or rivaroxaban in hip and knee replacement surgery: findings from the ORTHO-TEP registry. Thromb Haemost. 2013 Jan;109(1):154-63. doi: 10.1160/TH12-07-0510. Epub 2012 Nov 29. PMID 23197272
- [Background] Guyatt GH, Akl EA, Crowther M, Gutterman DD, Schuunemann HJ; American College of Chest Physicians Antithrombotic Therapy and Prevention of Thrombosis Panel. Executive summary: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):7S-47S. doi: 10.1378/chest.1412S3. No abstract available. PMID 22315257
- [Background] Lassen MR, Gent M, Kakkar AK, Eriksson BI, Homering M, Berkowitz SD, Turpie AG. The effects of rivaroxaban on the complications of surgery after total hip or knee replacement: results from the RECORD programme. J Bone Joint Surg Br. 2012 Nov;94(11):1573-8. doi: 10.1302/0301-620X.94B11.28955. PMID 23109641
- [Background] Granero J, Diaz de Rada P, Lozano LM, Martinez J, Herrera A; en nombre de los investigadores del grupo XAMOS Espana. [Rivaroxaban versus standard of care in venous thromboembolism prevention following hip or knee arthroplasty in daily clinical practice (Spanish data from the international study XAMOS)]. Rev Esp Cir Ortop Traumatol. 2016 Jan-Feb;60(1):44-52. doi: 10.1016/j.recot.2015.05.009. Epub 2015 Jul 17. Spanish. PMID 26194908
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03299296/Prot_SAP_001.pdf